CLINICAL TRIAL: NCT03500250
Title: Feasibility of a Nurse-led Intervention for the Early Management of Depression After Stroke in Hospital
Brief Title: Feasibility of the Post-Stroke Depression-toolkit
Status: Completed | Type: Observational
Sponsor: University of Applied Sciences Utrecht (Other)
Collaborators: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Dr. Mariska van Dijk, Dr., University of Applied Sciences Utrecht
Other Study IDs: PSD-toolkit
Record Dates: First submitted 2018-04-09; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Depression; Stroke
Keywords: Complex intervention; Depression; Nursing; Stroke; Feasibility
MeSH Terms: conditions — Depression; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nurses: Nurses working on the neurological wards of three hospitals (one university hospital and two general hospitals)
  Interventions: Other: Post-Stroke Depression toolkit

INTERVENTIONS:
Other: Post-Stroke Depression toolkit — The Post-Stroke Depression toolkit consists of three components: (1) two screening instruments, (2) seven evidence-based nursing interventions, and (3) an instruction manual.

SUMMARY:
Rationale: Depression is a frequent complication after a stroke. In stroke guidelines several recommendations focus on early screening, and treatment off depression after stroke. Introducing clinical practice guidelines into routine daily practice however, is a difficult process. In order to make the recommendations applicable to clinical practice a toolkit was developed (the Post Stroke Depression-toolkit), which provides assessment tools for the early detection of depression after stroke, and a set of interventions in case of a positive screening for (risk on) depressive symptoms.

Objective: to investigate the feasibility of the Post Stroke Depression-toolkit in daily practice.

Study design: An explanatory mixed-methods, before-and-after study design. Study population: Nurses working on the neurological wards of one university hospital and two general hospitals in the Netherlands were included in the study. Additionally, data were obtained from patient charts.

DETAILED DESCRIPTION:
Worldwide, approximately 50 million people who survived a stroke cope with physical, cognitive, and emotional impairments, and many of these survivors depend on caregivers to manage activities of daily living (Miller, et al., 2010). Stroke is the third leading cause of disability (Johnson, et al., 2016). Depression is a frequent and serious complication after stroke impeding rehabilitation outcome, and is associated with a higher mortality risk, and a lower quality of life (Kutlubaev & Hackett, 2014; Robinson & Jorge, 2015).

There is growing evidence for successful treatment of depression after stroke (Robinson & Jorge, 2015). Recommendations of stroke guidelines on the early management of depressive symptoms have not been structurally implemented in current practice, and only a minority of the acute care stroke teams assess mood on a systematic way in daily care (Hart & Bowen, 2008; Bowen, et al., 2005). Hence, depression is still one of the most underdiagnosed and undertreated complications after stroke (Miller et al., 2010), resulting in worse patient outcomes and delayed recovery (Robinson & Jorge, 2015). In a feasibility study of the Nursing Rehabilitation Guideline for Stroke (Hafsteinsdóttir & Schuurmans, 2009) it was suggested that simplifying the guideline and integrating the recommendations into a stroke care pathway could gain a more positive attitude towards the guideline and improve its feasibility (Hafsteinsdóttir et al., 2013). Therefore, the Post-Stroke Depression toolkit (PSD toolkit), an intervention for the early management of depression after stroke, has been developed.

The feasibility of this intervention was tested following phase two of the British Medical Research Council (MRC) guidelines (Craig et al., 2013). In this study, feasibility (Polit & Beck, 2008) is measured in terms of (1) fidelity, defined as the extent to which the components of the PSD toolkit are delivered as intended, and (2) acceptability, defined as whether the PSD toolkit is judged suitable and satisfactory by the nurses (Gearing et al., 2011). After evaluating implementation, the sustainability of the PSD toolkit requires evaluation as well (Scheirer, 2005). Sustainability is defined as fidelity to the PSD toolkit six months after completing implementation.

The aims of the study were (1) to explore the feasibility of the PSD toolkit in terms of fidelity and acceptability in three phases-a pre-implementation phase, an implementation phase, and a sustainability phase six month after-and (2) to identify elements for further refinement and improvement in the toolkit to enhance its feasibility in daily stroke care during the hospital stay.

Design: An explanatory mixed-methods, before-and-after study design(Creswell, 2008).

Data were collected by patient chart audits and surveys among nurses. Individual and focus group interviews with nurses followed the quantitative data collection to explain the findings (Creswell, 2008).

Data were collected pre-implementation in March and April 2012, during implementation from April 2012 until December 2012 and during the sustainability phase from December 2012 until June 2013.

A team with expertise in stroke care, consisting of two researchers and five nurses from the participating nursing teams, guided the implementation.

Participants and setting Nurses working on the neurological wards of one university hospital and two general hospitals in the Netherlands were included in the study. Additionally, data were obtained from patient charts.

Implementation strategies Evidence-based implementation strategies were used to facilitate the implementation of the PSD toolkit: (1) education and training of the nurses in applying the PSD toolkit, (2) opinion leaders, and (3) audit and feedback by the researcher (Van Achterberg et al., 2008).

Data collection Baseline data To gain insight into the patients in whom the toolkit was used, data on gender, age, marital status, living arrangements, type of stroke, length of hospital stay, and discharge destination were collected. The demographics collected on the nurses included gender, age, education, years working on the ward, and full-time equivalent.

Patient chart audit Fidelity was measured in terms of the extent to which the components of the PSD toolkit were applied as intended; patient chart audits were performed to establish the number of patients who were screened for depressive symptoms and who received nursing interventions in the case of a positive screening.

The Barriers and Facilitators Assessment Instrument To obtain a thorough understanding of the experiences and opinions of the nurses that influence fidelity, perceived barriers were evaluated using the Barriers and Facilitators Assessment Instrument (BFAI) (Peters et al., 2002)consisting of 18 statements, both positively and negatively formulated. One of the authors of the original questionnaire reviewed and approved the adaptations, confirming the content validity. The nurses indicated, on a five-point Likert scale, if they (dis)agreed with a statement. The scale ranged from 5 (strongly agree) to 1 (strongly disagree). To identify barriers, the percentage who agreed and strongly agreed with the positively formulated statements were recoded into disagree and strongly disagree; an item score of >3 (agree/strongly agree) indicating a barrier.

The Clinical Utility Questionnaire Acceptability was measured in terms of the clinical utility (Harris & Warren, 1995) of the PSD toolkit as perceived by the nurses. Clinical utility was assessed using an adapted version of the Clinical Utility Questionnaire including 19 items addressing nurses' views on the toolkit, focussing on item clarity, acceptability of time investment, utility of the instruments, and relevance and utility of the nursing interventions. The content validity of the adapted questionnaire was assessed by one of the authors of the original questionnaire (de Man-van Ginkel et al., 2012).

Interviews with nurses To explain the results of the audits, BFAI and the Clinical Utility Questionnaire, semi-structured with the nurses on the participating wards were performed at the end of the implementation phase and three focus group interviews were conducted at the end of the sustainability phase. The interview guides consisted of the following topics derived from results of the audits and questionnaires: (1) presentation of the quantitative results, (2) possible explanations for the changes (decrease/increase) in fidelity, (3) nurses' views on barriers or facilitators to use of the PSD toolkit and its clinical utility, and (4) suggestions to further improve the toolkit.

Procedure Pre-implementation phase Data was collected on daily nursing care regarding the management of depressive symptoms after stroke. The researchers examined the charts of all patients admitted to the participating wards using a data extraction form.

Furthermore, all nurses and nursing students received education and training sessions totalling three hours, which covered (1) depression after stroke (causes, consequences, and the importance of early detection of depressive symptoms), evidence-based nursing interventions, and (2) the content and procedures of the PSD toolkit.

Implementation phase The researcher visited the participating wards four times per week for patient chart audits to collect baseline data and data on fidelity of the PSD toolkit by registering the frequency of delivery of the components of the PSD toolkit by the nurses. The researchers sent the results of the patient chart audit (e.g., the proportion of patients who were screened for depressive symptoms and who received nursing interventions) to the opinion leaders. Subsequently, the opinion leaders used this overview to provide feedback and to remind the nurses to screen a patient for depressive symptoms and apply appropriate nursing interventions.

At the end of the implementation phase, the researchers sent the BFAI and Clinical Utility Questionnaire to the nurses. After two weeks, a reminder was sent to all non-respondents. Subsequently, the researchers conducted individual interviews with a random sample of five nurses from each of the participating nursing teams to explain fidelity to and acceptability of the toolkit by discussing the outcomes of the audit, the BFAI and the Clinical Utility Questionnaire.

Sustainability phase During the sustainability phase, the same procedure was used as in the implementation phase; however, no implementation strategies, such as feedback and reminders, were used by the opinion leaders. At the end of the sustainability phase, three explanatory focus group interviews (one with each team, consisting of 10, 12 and 6 participants) were conducted with a randomly selected group of nurses to explain the data on fidelity to and acceptability of the PSD toolkit. The focus group interviews were moderated by a researcher who was not involved in implementation. The researchers and the research assistants observed, took notes, and handled the recording devices.

Data analysis

* the baseline data, the audit data, and the results of the BFAI and Clinical Utility Questionnaire: Frequencies, means, standard deviations and percentages
* comparison of differences in patient groups: the Chi-square test for categorical baseline data and t-tests
* BFAI: numbers with the corresponding percentage of nurses who agreed and strongly agreed with an item on the questionnaire.
* the Clinical Utility Questionnaire: a percentage of agreement with each item.

A change of +/-10% in fidelity and acceptability was used to indicate an increase or decrease (McCluskey & Middleton, 2010). SPSS, version 23 (SPSS Inc., Chicago, IL, USA) was used for quantitative data analysis.

The individual and focus group interviews with the nurses were analysed according to predefined codes based on the topics in the interview guides. All interviews, as well as the focus groups, were audiotaped and transcribed verbatim. The transcripts were studied, and initial items were identified by a researcher, and subsequently, the items were discussed between two researchers. Based on consensus, the final items that explained the quantitative results on fidelity and acceptability of the PSD toolkit were established.

Ethical considerations This study received ethics approval from the Medical Ethics Committee of a University Medical Center (12-081C) and the local medical ethics committees of the participating hospitals. Informed consent was obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Registered Nurses with or without Bachelor degree in Nursing (BN); Nursing students.

Exclusion Criteria:

* none

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All nurses working on the neurological wards and stroke units of the participating hospitals, one university hospital and two general hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2013-06-30 (Actual); Study Completion 2013-06-30 (Actual)

PRIMARY OUTCOMES:
Fidelity | 12 months
  the extent to which the components of the PSD toolkit are delivered as intended
Acceptability | T=0; T=1 (after 6 months); T=2 (after 12 months)
  whether the PSD toolkit is judged suitable and satisfactory by the nurses

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M. Developing and evaluating complex interventions: the new Medical Research Council guidance. Int J Nurs Stud. 2013 May;50(5):587-92. doi: 10.1016/j.ijnurstu.2012.09.010. Epub 2012 Nov 15. No abstract available. PMID 23159157
- [Background] Research design: qualitative, quantitative and mixed methods approaches Research design: qualitative, quantitative and mixed methods approaches Creswell John W Sage 320 pound29 0761924426 0761924426 [Formula: see text]. Nurse Res. 2004 Sep 1;12(1):82-83. doi: 10.7748/nr.12.1.82.s2. PMID 28718745
- [Background] de Man-van Ginkel JM, Gooskens F, Schepers VP, Schuurmans MJ, Lindeman E, Hafsteinsdottir TB. Screening for poststroke depression using the patient health questionnaire. Nurs Res. 2012 Sep-Oct;61(5):333-41. doi: 10.1097/NNR.0b013e31825d9e9e. PMID 22710475
- [Background] Gearing RE, El-Bassel N, Ghesquiere A, Baldwin S, Gillies J, Ngeow E. Major ingredients of fidelity: a review and scientific guide to improving quality of intervention research implementation. Clin Psychol Rev. 2011 Feb;31(1):79-88. doi: 10.1016/j.cpr.2010.09.007. Epub 2010 Oct 7. PMID 21130938
- [Background] McCluskey A, Middleton S. Delivering an evidence-based outdoor journey intervention to people with stroke: barriers and enablers experienced by community rehabilitation teams. BMC Health Serv Res. 2010 Jan 19;10:18. doi: 10.1186/1472-6963-10-18. PMID 20082725
- [Background] Peters M., Harmsen M., Laurant M. & Wensing M. (2002) Barriers to and facilitators for improvement of patient care. Nijmegen: Centre for Quality of Care Research (WOK), Radboud University Nijmegen Medical Centre, the Netherlands.
- [Background] Polit, D. F., & Beck, C. T. (2008). Nursing research: Generating and assessing evidence for nursing practice Lippincott Williams & Wilkins.
- [Background] Scheirer, M. A. (2005). Is sustainability possible? A review and commentary on empirical studies of program sustainability. American Journal of Evaluation 26(3), 320-347.
- [Background] van Achterberg T, Schoonhoven L, Grol R. Nursing implementation science: how evidence-based nursing requires evidence-based implementation. J Nurs Scholarsh. 2008;40(4):302-10. doi: 10.1111/j.1547-5069.2008.00243.x. PMID 19094144
- [Background] Harris MR, Warren JJ. Patient outcomes: assessment issues for the CNS. Clin Nurse Spec. 1995 Mar;9(2):82-6. PMID 7600487
- [Background] Miller EL, Murray L, Richards L, Zorowitz RD, Bakas T, Clark P, Billinger SA; American Heart Association Council on Cardiovascular Nursing and the Stroke Council. Comprehensive overview of nursing and interdisciplinary rehabilitation care of the stroke patient: a scientific statement from the American Heart Association. Stroke. 2010 Oct;41(10):2402-48. doi: 10.1161/STR.0b013e3181e7512b. Epub 2010 Sep 2. No abstract available. PMID 20813995
- [Background] Johnson W, Onuma O, Owolabi M, Sachdev S. Stroke: a global response is needed. Bull World Health Organ. 2016 Sep 1;94(9):634-634A. doi: 10.2471/BLT.16.181636. No abstract available. PMID 27708464
- [Background] Kutlubaev MA, Hackett ML. Part II: predictors of depression after stroke and impact of depression on stroke outcome: an updated systematic review of observational studies. Int J Stroke. 2014 Dec;9(8):1026-36. doi: 10.1111/ijs.12356. Epub 2014 Aug 26. PMID 25156411
- [Background] Robinson RG, Jorge RE. Post-Stroke Depression: A Review. Am J Psychiatry. 2016 Mar 1;173(3):221-31. doi: 10.1176/appi.ajp.2015.15030363. Epub 2015 Dec 18. PMID 26684921
- [Background] Hart S, Morris R. Screening for depression after stroke: an exploration of professionals' compliance with guidelines. Clin Rehabil. 2008 Jan;22(1):60-70. doi: 10.1177/0269215507079841. Epub 2007 Nov 29. PMID 18048484
- [Background] Bowen A, Knapp P, Hoffman A, Lowe D. Psychological services for people with stroke: compliance with the U.K. National Clinical Guidelines. Clin Rehabil. 2005 May;19(3):323-30. doi: 10.1191/0269215505cr799oa. PMID 15859533
- [Background] Hafsteinsdottir TB, Varekamp R, Rensink M, van Linge R, Lindeman E, Schuurmans M; Rehabilitation Guideline Stroke Working Group. Feasibility of a nursing rehabilitation guideline for patients with stroke: evaluating the use by nurses. Disabil Rehabil. 2013 Jun;35(11):939-49. doi: 10.3109/09638288.2012.721049. Epub 2012 Oct 5. PMID 23035834
- [Background] Hafsteinsdóttir TB, Schuurmans MM. Clinical Nursing Rehabilitation Stroke-Guideline [in Dutch: Verpleegkundige Revalidatierichtlijn Beroerte. Maarsen: Elsevier Gezondheidszorg; 2009. Available from: http://www.elseviergezondheidszorg.nl
- [Derived] Van Dijk MJ, Hafsteinsdottir TB, Schuurmans MJ, de Man-van Ginkel JM. Feasibility of a nurse-led intervention for the early management of depression after stroke in hospital. J Adv Nurs. 2018 Dec;74(12):2882-2893. doi: 10.1111/jan.13806. Epub 2018 Aug 29. PMID 30019422